CLINICAL TRIAL: NCT05194540
Title: An Open-label, Single-arm, Phase 3 Trial to Evaluate the Efficacy and Safety of Tralokinumab Administered by an Autoinjector in Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: Efficacy and Safety of Tralokinumab Administered by an Autoinjector in Adults and Adolescents With Moderate to Severe Atopic Dermatitis (INJECZTRA)
Acronym: INJECZTRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0162-1338; U1111-1283-2072 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tralokinumab subcutaneous dosing by an autoinjector (Experimental): An initial SC dose of 600 mg tralokinumab at baseline followed by self-administration of a 300 mg dose of tralokinumab every other week for 14 weeks.
  Interventions: Drug: Tralokinumab

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of immunoglobulin G4 (IgG4) subclass that specifically binds to human interleukin-13 (IL-13) and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous administration

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of tralokinumab administered as subcutaneous (SC) injection by an autoinjector in adults and adolescents (age 12 to 17 years) with moderate-to-severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a single-arm, phase 3 trial designed to evaluate the efficacy and safety of tralokinumab when administered by an autoinjector in adults and adolescent subjects with moderate-to-severe AD. At baseline, the subjects will receive an initial SC dose of 600 mg tralokinumab. For the rest of the treatment period, all subjects will self-administer a dose of 300 mg tralokinumab every other week for 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years and above.
* Subject able and willing to self-administer tralokinumab with Device A.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD.
* History of AD for ≥1 year.
* A recent history (within 1 year before the screening visit) of inadequate response to treatment with topical medication or for whom topical treatments are otherwise medically inadvisable.
* AD involvement of ≥10% body surface area at screening and baseline.
* An EASI score of ≥12 at screening and ≥16 at baseline.
* An IGA score of ≥3 at screening and at baseline.
* Applied a stable dose of emollient twice daily (or more, as needed) for at least 14 days before baseline.

Exclusion Criteria:

* Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment.
* Use of tanning beds or phototherapy within 4 weeks prior to baseline.
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroids within 4 weeks prior to baseline.
* Treatment with topical corticosteroids, topical calcineurin inhibitors, topical phosphodiesterase 4 inhibitors, or topical Janus kinase inhibitors within 2 weeks prior to baseline.
* Receipt of any marketed biological therapy (i.e. immunoglobulin, anti immunoglobulin E) including dupilumab or investigational biologic agents 3 to 6 months prior to baseline.
* Active skin infections within 1 week prior to baseline.
* Clinically significant infection within 4 weeks prior to baseline.
* A helminth parasitic infection within 6 months prior to the date informed consent is obtained.
* Tuberculosis requiring treatment within 12 months prior to screening.
* Known primary immunodeficiency disorder.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (27):
- United States (27):
  - LEO Pharma Investigator, Birmingham, Alabama
  - LEO Pharma Investigator, Fort Smith, Arkansas
  - LEO Pharma Investigator, Fountain Valley, California
  - LEO Pharma Investigator, Fremont, California
  - LEO Pharma Investigational Site, Inglewood, California
  - LEO Pharma Investigator, Los Angeles, California
  - LEO Pharma Investigator, San Diego, California
  - LEO Pharma Investigator, Santa Ana, California
  - LEO Pharma Investigator, Centennial, Colorado
  - LEO Pharma Investigator, Farmington, Connecticut
  - LEO Pharma Investigational Site, Hialeah, Florida
  - LEO Pharma Investigator, Sanford, Florida
  - LEO Pharma Investigator, Libertyville, Illinois
  - LEO Pharma Investigator, Overland Park, Kansas
  - LEO Pharma Investigator, Bangor, Maine
  - LEO Pharma Investigator, Detroit, Michigan
  - LEO Pharma Investigator, Portsmouth, New Hampshire
  - LEO Pharma Investigator, Cortland, New York
  - LEO Pharma Investigator, Horseheads, New York
  - LEO Pharma Investigator, Bexley, Ohio
  - LEO Pharma Investigator, Toledo, Ohio
  - LEO Pharma Investigator, Tulsa, Oklahoma
  - LEO Pharma Investigator, Portland, Oregon
  - LEO Pharma Investigator, Dallas, Texas
  - LEO Pharma Investigator, Frisco, Texas
  - LEO Pharma Investigator, San Antonio, Texas
  - LEO Pharma Investigator, Webster, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soung J, Laquer V, Zirwas M, van Iperen P, Stinson JC, Albertsen KL, Stein Gold L. The Tralokinumab Pre-Filled Pen Improved Atopic Dermatitis Signs and Symptoms and Was Well Tolerated in Adults and Adolescents with Moderate-to-Severe Atopic Dermatitis: A 16-Week, Open-Label, Single-Arm Phase 3 Study (INJECZTRA). Dermatol Ther (Heidelb). 2025 Sep;15(9):2631-2644. doi: 10.1007/s13555-025-01490-3. Epub 2025 Jul 18. PMID 40681936

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tralokinumab Subcutaneous Dosing by an Autoinjector
Started | 136
Completed | 117
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Tralokinumab Subcutaneous Dosing by an Autoinjector
Number analyzed (Participants) | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 32
  White | 81
  More than one race | 5
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 136

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: IGA is an instrument used in clinical trials to rate the severity of the participant's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe)
Time Frame: At Week 16
Population: FAS, full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tralokinumab Subcutaneous Dosing by an Autoinjector
Number analyzed (Participants) | 136
percentage of subjects | 28.7 [21.7 to 36.8]

2. Primary Outcome: At Least 75% Reduction in Eczema Area and Severity Index (EASI75) at Week 16
Description: Eczema Area and Severity Index (EASI) is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. EASI is a composite index with scores ranging from 0 to 72, where higher values indicate a more severe or more extensive condition
Time Frame: At Week 16
Population: FAS, full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tralokinumab Subcutaneous Dosing by an Autoinjector
Number analyzed (Participants) | 136
percentage of subjects | 43.4 [35.3 to 51.8]

3. Secondary Outcome: Number of Treatment-emergent Adverse Events (AEs) From Baseline to Week 16
Description: An AE will be considered treatment emergent if it started after the first injection of trial drug
Time Frame: From Week 0 to Week 16
Population: SAF, safety analysis set
Measure: Number; unit: events
Arm/Group | Tralokinumab Subcutaneous Dosing by an Autoinjector
Number analyzed (Participants) | 136
events | 86

4. Secondary Outcome: Presence of Treatment-emergent Anti-drug Antibodies (ADA) From Baseline to Week 16
Description: Serum samples for determination of presence or absence of ADA will be analysed using a validated bioanalytical method
Time Frame: From Week 0 to Week 16
Population: SAF, safety analysis set
Measure: Number; unit: participants
Arm/Group | Tralokinumab Subcutaneous Dosing by an Autoinjector
Number analyzed (Participants) | 136
participants | 0

ADVERSE EVENTS:
Time Frame: Initial Treatment Period: Week 0 to week 16, Safety Follow- Up Period: Week 16 to Week 20.
Groups:
- Tralokinumab+TCS Initial Treatment Period Week 0 to Week 16: Tralokinumab+TCS (N=136)
- Safety Follow-Up Week 16 to Week 20: Safety Follow-Up (N=131)
Arm/Group | Tralokinumab+TCS Initial Treatment Period Week 0 to Week 16 | Safety Follow-Up Week 16 to Week 20
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/131
Other Adverse Events (participants affected / at risk) | 24/136 | 0/131
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab+TCS Initial Treatment Period Week 0 to Week 16 (N=136) | Safety Follow-Up Week 16 to Week 20 (N=131)
Injection site pain (General disorders) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 8 (10) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (4) | 0 (0)
Dermatitis infected (Infections and infestations) | 3 (3) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT05194540/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT05194540/SAP_001.pdf